CLINICAL TRIAL: NCT04843696
Title: Negative Pressure Ventilation-rehabilitation on Acute Exacerbation and Associated Molecular Biomarkers and Cytokines in Chronic Obstructive Pulmonary Disease Over 2 Years
Brief Title: Negative Pressure Ventilation-rehabilitation on Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902168B0
Record Dates: First submitted 2021-04-06; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Acute Exacerbation of COPD
Keywords: Chronic obstructive pulmonary disease; Negative-pressure ventilation; Acute Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPV group (Experimental): The hospital-based maintenance NPV program includes NPV support, breathing training, and an educational program (relaxation techniques and a home pacing walking exercise) in daily clinical practice. The patients in the NPV group undergo the hospital-based NPV once per week in the maintenance program at least three times per month.
  The patients received NPV with breathing training via a cuirass ventilator (cuirass diameter 21 cm or 34 cm, Dima Italia Srl.,Bologna, Italy) for 60 min, once per week.
  Breathing training consisted of breathing techniques (pursued-lipped, controlled, and diaphragmatic breathing).
  Interventions: Device: cuirass ventilator (cuirass diameter 21 cm or 34 cm, Dima Italia Srl.,Bologna, Italy); Behavioral: breathing training, and an educational program (relaxation techniques and a home pacing walking exercise)
- Control group (Active Comparator): Control group receives breathing training, and an educational program (relaxation techniques and a home pacing walking exercise) in daily clinical practice.
  Breathing training consisted of breathing techniques (pursued-lipped, controlled, and diaphragmatic breathing).
  Interventions: Behavioral: breathing training, and an educational program (relaxation techniques and a home pacing walking exercise)

INTERVENTIONS:
Device: cuirass ventilator (cuirass diameter 21 cm or 34 cm, Dima Italia Srl.,Bologna, Italy) — the hospital-based NPV once per week in the maintenance program at least three times per month. The ventilator is set to the control model with a frequency of 12~15 cycles/min, 30% of the ratio of inspiratory time to total breathing cycle time (Ti/Ttot), and delivery of negative pressures ranging from -20 to -35 cm H2O.
  Arms: NPV group
Behavioral: breathing training, and an educational program (relaxation techniques and a home pacing walking exercise) — breathing training, and an educational program (relaxation techniques and a home pacing walking exercise) Breathing training consisted of breathing techniques (pursued-lipped, controlled, and diaphragmatic breathing)

SUMMARY:
This investigator-initiated, prospective, single center, randomized, controlled clinical trial enrolled patients with stable Global Initiative for Chronic Obstructive Lung Disease stage II-IV chronic obstruction pulmonary disease. The primary outcome was 2-year acute exacerbation rates.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR) has been suggested to be positive effects on 6 min walking distance (6MWD), muscle force, cycle exercise endurance time, and quality of life. However, the literature still could not explain the role of PR in reducing systemic inflammation of chronic obstruction pulmonary disease (COPD) patients. A recent study found that PR with negative pressure ventilation (NPV) improved lung function, exercise capacity and reduced acute exacerbation rates in COPD patients. The objectives of this research are to design a prospective, randomized controlled trial to determine the clinical outcome of NPV-PR in COPD patients and to investigate if NPV-PR reduces systemic inflammation in patients with COPD.

This investigator-initiated, prospective, single center, randomized, controlled clinical trial enrolled patients with stable Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage II-IV COPD. NPV was targeted to reduce baseline blood carbon dioxide by at least 20% during NPV titration. Patients were randomly assigned (in a 1:1 ratio) to continue optimised standard treatment (control group) or to receive additional NPV-PR for at least 24 months (intervention group). The primary outcome was 2-year acute exacerbation rates. The lung function and walking distance will be assessed by six-minute walking tests and the severity of disease will be evaluated by high resolution computed tomography scores. Peripheral blood sample will be collected to analyze the inflammatory cytokines and oxidative markers.

In the present prospective study, investigators hypothesize that NPV-PR would be superior to usual care in reducing the risk for acute exacerbations of COPD, hospitalisations and emergency visits over a 24-month period. This research will provide evidence for the role of NPV-PR in the management of COPD, and evidence for a role of systemic inflammation in disease progression of COPD. The results may provide certain insights into more effective treatments to inhibit the disease progression of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD ((post-bronchodilation forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC) <0.7)
* Optimal medical treatment according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD)) at least 3 months before screening

Exclusion Criteria:

* abnormalities of the thorax or the lung other than COPD,
* acute exacerbation within one month
* obesity with a body-mass index (BMI) ≥35 kg/m²,
* malignant co-morbidities, severe heart failure (New York Heart Association stage IV), unstable angina, severe arrhythmias, neuromuscular diseases and/or impairment of basal brain nerve function with disturbed swallowing and choking and impaired general condition that could preclude regular follow-up visits.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
COPD acute exacerbations rate | 2 years
  mild (required treatment with oral/systemic corticosteroids and/or antibiotics, without hospitalization) moderate (required treatment with oral/systemic corticosteroids and/or antibiotics, with emergency department visits) severe (required in-patient hospitalization)

SECONDARY OUTCOMES:
the yearly rate of decline of forced expiratory volume in 1 second (FEV1) | 2 years
  the yearly rate of decline of FEV1
the yearly rate of decline of 6 minute walking distance (6MWD) | 2 years
  the yearly rate of decline of 6MWD
Mortality | 2 years
  overall and pulmonary related

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
The IRB of Chang Gung Memorial Hospital does not permit to share IPD in this project.

REFERENCES:
- [Background] Huang HY, Lo CY, Yang LY, Chung FT, Sheng TF, Lin HC, Lin CW, Huang YC, Chang CJ, Chung KF, Wang CH. Maintenance Negative Pressure Ventilation Improves Survival in COPD Patients with Exercise Desaturation. J Clin Med. 2019 Apr 25;8(4):562. doi: 10.3390/jcm8040562. PMID 31027263
- [Background] Huang HY, Chou PC, Joa WC, Chen LF, Sheng TF, Lin HC, Yang LY, Pan YB, Chung FT, Wang CH, Kuo HP. Pulmonary rehabilitation coupled with negative pressure ventilation decreases decline in lung function, hospitalizations, and medical cost in COPD: A 5-year study. Medicine (Baltimore). 2016 Oct;95(41):e5119. doi: 10.1097/MD.0000000000005119. PMID 27741132